CLINICAL TRIAL: NCT06691802
Title: Clinical Study on Reducing Recurrent Attacks of Chronic Airway Diseases (asthma, Chronic Obstructive Pulmonary Disease) with Shu Fei Tie Based on "winter Disease Being Cared in Summer"
Brief Title: Clinical Study on the Treatment of Chronic Airway Diseases (Asthma, Chronic Obstructive Pulmonary Disease) with Shu Fei Tie
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Qingdao Municipal Hospital of Traditional Chinese Medicine (Unknown); Henan Lingrui Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chronic Airway Diseases
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmoriary Disease (COPD); Asthma
Keywords: Chronic Obstructive Pulmoriary Disease; Asthma; Shu Fei Tie; Winter disease being cared in summer; Randomized Controlled Trial
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shu Fei Tie group for Asthma/COPD (Experimental): Patients in the Asthma/COPD experimental group were treated with Shu Fei Tie
  Interventions: Drug: Shu Fei Tie
- Shu Fei Tie Placebo group for Asthma/COPD (Placebo Comparator): Patients in the Asthma/COPD experimental group were treated with Shu Fei Tie Placebo
  Interventions: Drug: Shu Fei Tie placebo

INTERVENTIONS:
Drug: Shu Fei Tie — Optimize the extraction process and matrix formulation, and combine the use of traditional Chinese medicine volatile oil and chemical transdermal enhancers to develop adermal patch（Shu Fei Tie）
  Arms: Shu Fei Tie group for Asthma/COPD
Drug: Shu Fei Tie placebo — Shu Fei Tie Placebos are made using substances without active drug ingredients, following the same preparation procedures
  Arms: Shu Fei Tie Placebo group for Asthma/COPD

SUMMARY:
Conduct a multi-center, large-sample, randomized controlled clinical study of "winter disease being cared in summer" with Shu Fei Tie prevent recurrence of Asthma and COPD, scientifically evaluate the clinical efficacy and safety of Shu Fei Tie in reducing the recurrence of chronic airway diseases, identify target population, clarify the mechanism of efficacy, and establish a prevention and treatment technology plan for Shu Fei Tie to reduce the recurrence of chronic airway diseases.

DETAILED DESCRIPTION:
Asthma and Chronic obstructive pulmonary disease (COPD) are the most common chronic airway diseases, and their recurrent episodes or acute exacerbations are the main reasons for the decline in patients' quality of life and heavy economic burden. Based on the of "winter disease being cared in summer", traditional Chinese medicine (TCM) has a long history and wide application in preventing and treating the recurrence of chronic air diseases, with obvious advantages of combining TCM and Western medicine. However, there is a lack of integrated TCM and Western medicine technical schemes for chronic airway based on high-level evidence-based evidence. The Shu Fei Tie developed by our project team is a medical institution preparation that has been used clinically for a long. Therefore, this study conducted a multi-center, large-sample, randomized controlled clinical study of the Shu Fei Tie to prevent the recurrence of asthma and COPD. The study subjects were patients in the remission period of asthma (1332 cases) and the stable period of COPD (980 cases) On the basis of treatment guided by the guidelines, the experimental group was given the Shu Fei Tie, and the control group was given a placebo of theu Fei Tie. The treatment started 10 days before the " the first Fu" and was conducted every 10 days, A total of 5 times, Each treatment lasted 6-8 hours, and the follow-up period was 45 weeks, for a total of 3 cycles (3 years). The outcome indicators were the number of acute attacks per year for asthma and the number of acute exacerbations per year for COPD. The secondary outcome indicators for asthma included Asthma Control Test (ACT) score, the Asthma Control Questionnaire (ACQ), and the Asthma Quality of Life Questionnaire (AQLQ). For COPD, the secondary outcome indicators included clinical symptom scores and lung function. This study scientifically evaluated the clinical efficacy and safety of the Shu Fei Tie reducing the recurrence of chronic airway diseases, identified the advantageous population, elucidated the mechanism of efficacy, and established a technical scheme for preventing and treating the recurrence of chronic airway diseases with the Shu Fei Tie.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for asthma/COPD(Group E in the GOLD classification); ② Age range from18 years to 80 years(asthma) and 40 yesrs to 80 years(COPD);

  * The investigators agreed to participate in this clinical study by voluntarily signing an informed consent form.

Exclusion Criteria:

* Patients with other pulmonary diseases (lung abscess, pulmonary interstitial fibrosis, active pulmonary tuberculosis, bronchiectasis，etc);

  * Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina, acute myocardial infarction, heart grade 3 or above, stroke, cerebral hemorrhage, etc.);

    * Patients with severe liver diseases (liver cirrhosis, portal hypertension, and caused by esophageal and gastric varices) and severe kidney diseases (dialysis, kidney transplantation, etc.);

      * Patients with impaired consciousness or various illnesses who cannot communicate normally; ⑤Pregnant and lactating women; ⑥Patients who are participating in other clinical trials within one month prior to enrollment; ⑦Patients who have received acupuncture or other traditional Chinese medicine external treatments within the past year; ⑧ Patients who are allergic to external patches

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2312 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Asthma part：Number of acute attacks per year | Count once a year for three consecutive years
  Record the number of acute attacks per year for each patient, and evaluate the effect of the lung-clearing patch on reducing the number of acute attacks
COPD part：The number of acute exacerbations per year | Count once a year for three consecutive years
  Record the number of acute exacerbations in patients per year to evaluate the treatment effect of Shu Fei Tie on patients.
COPD part：the interval between successive acute exacerbations | at weeks 13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)，Until the first acute exacerbation occurs
  Record relevant information and evaluate the treatment effect of lung soothing patches on patients.
COPD part:the number of rehospitalizations within a year | Count once a year until the end of the 3-year cycle
  Record relevant information and evaluate the treatment effect of lung soothing patches on patients.

SECONDARY OUTCOMES:
Asthma part：Asthma Control Test | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  ACT includes five questions. Every question will be assessed using a 5-point scale with scores ranging from 5 to 25. The higher the score, the better the symptom control.25 is considered complete control level, 20 ~ 24 is considered good control level, and <20 is considered non-control level.
Asthma part：Asthma Control Questionnaire | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  The content of ACQ involves the following aspects: asthma-related, symptoms, the use of first-aid drugs, the impact on daily life and lung function test results.The higher the score, the worse the state.
Asthma part：Asthma Quality of Life Questionnaire | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  The asthma quality of life scale (5-point scale-RRB- consists of 35 items, including activity limitation (1-12) , asthma symptoms (13-20) , psychological status (22-26) , response to stimuli (27-31) , concern for one's own health (32-35) . On a 5-point scale, 1 is the worst and 5 is the best.
Asthma part：Frequency of anti-inflammatory and analgesic use | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  Detailed record of the use of treatment drugs, evaluation of treatment effect
Asthma part：Disease Control Rate | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  Based on the disease control situation, the disease control rate is calculated and the efficacy is evaluated.
Asthma part：readmission rate | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  The impact on patient prognosis was evaluated by calculating the number of readmissions.
Asthma part：Forced expiratory volume in the first second | Before treatment, at weeks 52, 104, and 156 of treatment
  FEV1 will be applied to assess pulmonary function
Asthma part：Peak expiratory flow | Before treatment, at weeks 52, 104, and 156 of treatment
  PEF will be applied to assess pulmonary function
Asthma part：Fractional exhaled nitric oxide | Before treatment, at weeks 52, 104, and 156 of treatment
  PEF will be used to evaluate the patient's airway inflammation
Asthma part：clinical symptoms and signs questionnaire | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, expectoration, chest tightness, gasp and wheezing. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
COPD part：clinical symptoms and signs questionnaire | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, phlegm, chest tightness, gasp,shortness of breath, feeble and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
COPD part：mMRC | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
COPD part：CAT | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  0-40 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was >10, the participant needed to be seen by a physician for further testing to determine if they had COPD.
COPD part：SGRQ | at weeks 0,13, 26, 39, and 52, for 3 consecutive cycles (each cycle is 1 year)
  The evaluation content consists of three parts: respiratory symptoms, activity ability, and disease impact. The questionnaire is calculated using SGRQ software, and the symptom score, activity score, impact score, and total score are obtained separately. The score fluctuates between 0-100, and the quality of life is negatively correlated with the score.
COPD part：Forced expiratory volume in the first second | Before treatment, at weeks 52, 104, and 156 of treatment
  FEV1 will be applied to assess pulmonary function
COPD part：Forced Vital Capacity | Before treatment, at weeks 52, 104, and 156 of treatment
  FVC will be applied to assess pulmonary function
COPD part：Forced expiratory volume in the first Second Percentage of predicted value | Before treatment, at weeks 52, 104, and 156 of treatment
  FEV1% will be applied to assess pulmonary function
COPD part：Maximal Mid-Expiratory Flow | Before treatment, at weeks 52, 104, and 156 of treatment
  MMEF will be applied to assess pulmonary function
COPD part：Forced expiratory flow at 50% of FVC exhaled | Before treatment, at weeks 52, 104, and 156 of treatment
  FEF50% will be applied to assess pulmonary function
COPD part：Forced expiratory flow at 75% of FVC exhaled | Before treatment, at weeks 52, 104, and 156 of treatment
  FEF75% will be applied to assess pulmonary function

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China